CLINICAL TRIAL: NCT05874115
Title: Development of a Biomarker to Predict the Efficacy of Anti-angiogenic Therapy in Ovarian Cancer
Acronym: OutCoME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO2019.053
Record Dates: First submitted 2023-04-26; First posted 2023-05-24 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: liquid biopsy — liquid biopsy

SUMMARY:
Epithelial ovarian cancer (EOC) is a highly angiogenic tumor and drug targeting of angiogenesis is effective in some selected groups of EOC patients. However, no biomarkers are available to predict the effectiveness of this expensive therapy.Investigators believe that Multimerin-2, an extracellular matrix molecule, could serve as a biomarker that can address this clinical need. Multimerin-2 is deposited throughout the vasculature and its expression in EOC-associated vessels is frequently lost, in part due to increased degradation. Multimerin-2 sequesters VEGFA and other angiogenic factors and their release upon degradation of Multimerin-2 could underlie resistance to anti-angiogenic therapy. Indeed, fragments of degradation of Multimerin-2 are found in high concentrations in sera of EOC patients. Furthermore, the loss of Multimerin-2 impairs the function of the vessels, and this could negatively affect the delivery of the drug and the efficacy of the treatment.

With the aim of predicting the efficiency of anti-angiogenic therapy, researchers will evaluate the angiogenic properties and expression of Multimerin-2 in EOC tumors, and develop a new Multimerin-2-based biomarker detectable by liquid biopsy, in order to manage EOC patients in a targeted manner based on the biological characteristics of their tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years
2. Histological diagnosis of epithelial carcinoma of the ovary or fallopian tubes or primary carcinoma of the peritoneum, including mixed Mullerian tumours.
3. Stage IIIb, IIIc or IV
4. Performance Status 0-2 according to ECOG
5. Availability of tumor tissue samples and biological fluids for molecular analyses
6. Informed consent for the collection, storage and use of biological material for the CRO Biobank (as specified in the consent of the CRO Biobank, Rev 2 of 03/10/2016), signed and obtained before surgery for suspected EOC.

Exclusion Criteria:

1. Ovarian tumors of low malignant potential (i.e. borderline tumors)
2. Other malignacies within the last 5 years except carcinoma in situ of the cervix or early stage squamous cell or basal cell carcinoma of the skin, as long as they are adequately treated.
3. Active infection or uncontrolled chronic inflammatory disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with histological diagnosis of epithelial ovarian carcinoma (EOC),consecutively referred to the IRCCS CRO of Aviano in the study period
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Multimerin-2 levels and progression free survival | from EOC diagnosis diagnosis until first documented progression or death from any cause, up to 2 years
  To investigate whether Multimerin-2 level measured in serum could represent a potential prognostic biomarker (measured as progression free survival) in bevacizumab-treated subjects
Multimerin-2 levels and progression free survival | from EOC diagnosis diagnosis until first documented progression or death from any cause, up to 2 years
  To investigate whether Multimerin-2 level measured in urine could represent a potential prognostic biomarker (measured as progression free survival) in bevacizumab-treated subjects
Multimerin-2 levels and progression free survival | from EOC diagnosis diagnosis until first documented progression or death from any cause, up to 2 years
  To investigate whether Multimerin-2 level measured in ascites could represent a potential prognostic biomarker (measured as progression free survival) in bevacizumab-treated subjects

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Maurizio, Principal Investigator — Centro di Riferimento Oncologico (CRO), IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO), IRCCS, Aviano, Italy

IPD SHARING:
Plan to Share IPD: No